CLINICAL TRIAL: NCT05282108
Title: Efficacy and Safety of Generic Imatinib (Carcemia®) Compared to Glivec® in Real-Life Management of Chronic Phase of Chronic Myeloid Leukemia; a Multicenter, Observational Study
Brief Title: Efficacy and Safety of Generic Imatinib (Carcemia®) Compared to Glivec® in Real-Life Management of Chronic Phase of Chronic Myeloid Leukemia
Acronym: CARCML
Status: Recruiting | Type: Observational
Sponsor: Hikma Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: HIK-CAR-2021-04
Record Dates: First submitted 2022-03-03; First posted 2022-03-16 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Imatinib; Carcemia; Leukemia; Cohort study; Effectiveness; Safety; Observational study; Cancer; Blood cancer; Health related qulaity of life; Glivec
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia; Neoplasms; Hematologic Neoplasms | interventions — Imatinib Mesylate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Carcemia group: The cohort treated with Carcemia
  Interventions: Drug: Carcemia
- Glivec Group: The cohort treated with Glivec
  Interventions: Drug: Glivec

INTERVENTIONS:
Drug: Carcemia — Generic Imatinib
  Groups: Carcemia group
Drug: Glivec — Imatinib
  Groups: Glivec Group

SUMMARY:
The purpose of this study is to evaluate Efficacy and Safety of Generic Imatinib (Carcemia®) Compared to Glivec® in Real-Life Management of Chronic Phase of Chronic Myeloid Leukemia

DETAILED DESCRIPTION:
This is an observational, prospective, cohort study design, where no visits or intervention(s) additional to the daily practice will be performed. In the study site, two cohorts will be identified among eligible patients, followed up, and assessed for a total of 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Newly diagnosed patients with Ph+ CML in CP, with or without the presence of other cytogenetic abnormalities at the time of diagnosis
3. Treatment naïve patients with confirmed diagnosis within 3 months of study enrolment
4. Levels of liver aminotransferases and serum bilirubin ≤ 2 times the upper limit of the normal range, and serum creatinine ≤1.5 times the upper limit of the normal range
5. Written informed consent

Exclusion Criteria:

1. CML in accelerated phase (AP) at enrolment except patients in AP with the presence of other cytogenetic abnormalities at the time of diagnosis 2. CML in BP at enrolment 3. Patients who meet any of the contraindications to the administration of the study drug according to the approved Summary of Product Characteristics.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from different sites in Egypt
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who achieve and maintain major molecular response (MMR) at 12 months | 12 months
  Proportion of patients who achieve and maintain major molecular response (MMR) at 12 months using RQ-PCR test (Appendix II) using Chi-square test. The MMR is defined as ration of BCR-ABL to ABL (or other housekeeping gene) ≤ 0.1% on the international scale (MMR is equal to a 3-log reduction in the ratio of BCR-ABL1: ABL from a standardized median baseline value).

SECONDARY OUTCOMES:
the safety & tolerability of imatinib after 12 months | 12 months
  In both cohorts, the safety & tolerability of imatinib after 12 months of treatment will be assessed by:
  * The number, type, severity and frequency of the adverse reactions particularly those described in the SmPC of the reference product.
  * Incidence of adverse events (AEs) & serious adverse events (SAEs).
  * AEs leading to permanent treatment discontinuation.
  * Clinically relevant changes in laboratory tests (according to laboratory reference ranges).
Progression free survival (PFS) at 12 months | 12 months
Event free survival (EFS) at 12 months | 12 months
Survival without blastic phase (BP) at 12 months | 12 months
Overall survival (OS) at 12 months | 12 months
Complete cytogenetic response (CCyR) at 12 months | 12 months
Deep Molecular response (DMR) at 12 months | 12 months
Treatment compliance | 12 months
  Treatment compliance while on imatinib will be evaluated by identifying the frequency of not taking the medications as prescribed and the reason behind that based on the prescription pattern. The decision on non-compliance is based on the treating physician's judgment."

CONTACTS AND LOCATIONS:
Locations (4):
- Egypt (4):
  - National Cancer Institute (NCI), Cairo
  - Ain Shams University Hospital, Cairo
  - Nasser Institute, Cairo
  - Tanta Oncology Center, Tanta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ercaliskan A, Seyhan Erdogan D, Eskazan AE. Current evidence on the efficacy and safety of generic imatinib in CML and the impact of generics on health care costs. Blood Adv. 2021 Sep 14;5(17):3344-3353. doi: 10.1182/bloodadvances.2021004194. PMID 34477815
- [Background] Abou Dalle I, Kantarjian H, Burger J, Estrov Z, Ohanian M, Verstovsek S, Ravandi F, Borthakur G, Garcia-Manero G, Jabbour E, Cortes J. Efficacy and safety of generic imatinib after switching from original imatinib in patients treated for chronic myeloid leukemia in the United States. Cancer Med. 2019 Nov;8(15):6559-6565. doi: 10.1002/cam4.2545. Epub 2019 Sep 10. PMID 31502383
- [Background] Awidi A, Abbasi S, Alrabi K, Kheirallah KA. Generic Imatinib Therapy Among Jordanians: An Observational Assessment of Efficacy and Safety in Routine Clinical Practice. Clin Lymphoma Myeloma Leuk. 2017 Dec;17(12):e55-e61. doi: 10.1016/j.clml.2017.08.001. Epub 2017 Aug 5. PMID 28844599
- [Background] Danthala M, Gundeti S, Kuruva SP, Puligundla KC, Adusumilli P, Karnam AP, Bala S, Konatam ML, Maddali LS, Digumarti RR. Generic Imatinib in Chronic Myeloid Leukemia: Survival of the Cheapest. Clin Lymphoma Myeloma Leuk. 2017 Jul;17(7):457-462. doi: 10.1016/j.clml.2017.05.006. Epub 2017 May 10. PMID 28559151
- [Background] Jiang H, Zhi LT, Hou M, Wang JX, Wu DP, Huang XJ. [Comparison of generic and original imatinib in the treatment of newly diagnosed patients with chronic myelogenous leukemia in chronic phase: a multicenter retrospective clinical study]. Zhonghua Xue Ye Xue Za Zhi. 2017 Jul 14;38(7):566-571. doi: 10.3760/cma.j.issn.0253-2727.2017.07.003. Chinese. PMID 28810322
- [Background] Gemelli M, Elli EM, Elena C, Iurlo A, Intermesoli T, Maffioli M, Pungolino E, Carraro MC, D'Adda M, Lunghi F, Anghileri M, Polverelli N, Rossi M, Bacciocchi M, Bono E, Bucelli C, Passamonti F, Antolini L, Gambacorti-Passerini C. Use of generic imatinib as first-line treatment in patients with chronic myeloid leukemia (CML): the GIMS (Glivec to Imatinib Switch) study. Blood Res. 2020 Sep 30;55(3):139-145. doi: 10.5045/br.2020.2020130. PMID 32792470
- [Background] Deininger MW, Shah NP, Altman JK, Berman E, Bhatia R, Bhatnagar B, DeAngelo DJ, Gotlib J, Hobbs G, Maness L, Mead M, Metheny L, Mohan S, Moore JO, Naqvi K, Oehler V, Pallera AM, Patnaik M, Pratz K, Pusic I, Rose MG, Smith BD, Snyder DS, Sweet KL, Talpaz M, Thompson J, Yang DT, Gregory KM, Sundar H. Chronic Myeloid Leukemia, Version 2.2021, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2020 Oct 1;18(10):1385-1415. doi: 10.6004/jnccn.2020.0047. PMID 33022644
- [Background] Jabbour E, Kantarjian H. Chronic myeloid leukemia: 2016 update on diagnosis, therapy, and monitoring. Am J Hematol. 2016 Feb;91(2):252-65. doi: 10.1002/ajh.24275. PMID 26799612
- [Background] Baccarani M, Cortes J, Pane F, Niederwieser D, Saglio G, Apperley J, Cervantes F, Deininger M, Gratwohl A, Guilhot F, Hochhaus A, Horowitz M, Hughes T, Kantarjian H, Larson R, Radich J, Simonsson B, Silver RT, Goldman J, Hehlmann R; European LeukemiaNet. Chronic myeloid leukemia: an update of concepts and management recommendations of European LeukemiaNet. J Clin Oncol. 2009 Dec 10;27(35):6041-51. doi: 10.1200/JCO.2009.25.0779. Epub 2009 Nov 2. PMID 19884523
- [Background] Baccarani M, Deininger MW, Rosti G, Hochhaus A, Soverini S, Apperley JF, Cervantes F, Clark RE, Cortes JE, Guilhot F, Hjorth-Hansen H, Hughes TP, Kantarjian HM, Kim DW, Larson RA, Lipton JH, Mahon FX, Martinelli G, Mayer J, Muller MC, Niederwieser D, Pane F, Radich JP, Rousselot P, Saglio G, Saussele S, Schiffer C, Silver R, Simonsson B, Steegmann JL, Goldman JM, Hehlmann R. European LeukemiaNet recommendations for the management of chronic myeloid leukemia: 2013. Blood. 2013 Aug 8;122(6):872-84. doi: 10.1182/blood-2013-05-501569. Epub 2013 Jun 26. PMID 23803709
- [Background] Hochhaus A, Baccarani M, Silver RT, Schiffer C, Apperley JF, Cervantes F, Clark RE, Cortes JE, Deininger MW, Guilhot F, Hjorth-Hansen H, Hughes TP, Janssen JJWM, Kantarjian HM, Kim DW, Larson RA, Lipton JH, Mahon FX, Mayer J, Nicolini F, Niederwieser D, Pane F, Radich JP, Rea D, Richter J, Rosti G, Rousselot P, Saglio G, Saussele S, Soverini S, Steegmann JL, Turkina A, Zaritskey A, Hehlmann R. European LeukemiaNet 2020 recommendations for treating chronic myeloid leukemia. Leukemia. 2020 Apr;34(4):966-984. doi: 10.1038/s41375-020-0776-2. Epub 2020 Mar 3. PMID 32127639
- [Background] O'Brien SG, Guilhot F, Larson RA, Gathmann I, Baccarani M, Cervantes F, Cornelissen JJ, Fischer T, Hochhaus A, Hughes T, Lechner K, Nielsen JL, Rousselot P, Reiffers J, Saglio G, Shepherd J, Simonsson B, Gratwohl A, Goldman JM, Kantarjian H, Taylor K, Verhoef G, Bolton AE, Capdeville R, Druker BJ; IRIS Investigators. Imatinib compared with interferon and low-dose cytarabine for newly diagnosed chronic-phase chronic myeloid leukemia. N Engl J Med. 2003 Mar 13;348(11):994-1004. doi: 10.1056/NEJMoa022457. PMID 12637609
- [Background] Kantarjian H, O'Brien S, Jabbour E, Shan J, Ravandi F, Kadia T, Faderl S, Garcia-Manero G, Borthakur G, Cortes J. Impact of treatment end point definitions on perceived differences in long-term outcome with tyrosine kinase inhibitor therapy in chronic myeloid leukemia. J Clin Oncol. 2011 Aug 10;29(23):3173-8. doi: 10.1200/JCO.2010.33.4169. Epub 2011 Jul 11. PMID 21747082
- [Background] Deininger MW, O'Brien SG, Ford JM, Druker BJ. Practical management of patients with chronic myeloid leukemia receiving imatinib. J Clin Oncol. 2003 Apr 15;21(8):1637-47. doi: 10.1200/JCO.2003.11.143. Epub 2003 Mar 13. PMID 12668652